CLINICAL TRIAL: NCT05963360
Title: Planning for Frailty: Optimal Health and Social Care Workforce Organisation Using Demand-led Simulation Modelling (FLOWS)
Brief Title: Planning for Frailty: Optimal Health and Social Care Workforce Organisation Using Demand-led Simulation Modelling
Acronym: FLOWS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Bournemouth University (Other); Tameside Hospital NHS Foundation Trust (Other); Southern Health NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 71937
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Frailty in Aging; Older People
Keywords: Planning for Frailty; Health and Social Care Workforce Organisation; Social care Workforce; Simulation Modelling; Health Workforce

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Frailty in Older people: Older people, 50 and above.

SUMMARY:
What is the present, and expected, size and composition of the health and social care workforce required to provide care for the frail older population? As the population ages, robust workforce planning to meet future demands for health and social care by older people is needed. A lack of evidence in this areas has led to a mis-match between the health and social care demand from the ageing population and the current workforce capacity. The proposed study will use demand-led simulation modelling of the workforce required to address the specific challenge of providing health and social care for the growing numbers of older people living with frailty.

DETAILED DESCRIPTION:
Research Question: What is the present, and expected, size and composition of the health and social care workforce required to provide care for the frail older population? Background: As the population ages, robust workforce planning to meet future demands for health and social care by older people is needed. A lack of evidence in this area has led to a mis-match between the health and social care demand from the ageing population and the current workforce capacity. The proposed study will use demand-led simulation modelling of the workforce required to address the specific challenge of providing health and social care for the growing numbers of older people living with frailty.

Aims & Objectives: The aim of the study is to use simulation modelling to explore long-term trends in frailty-related health and social care use in the ageing population and its implications for future workforce size and competencies to support high quality care. The primary objective of this study is the creation of a simulation model that will inform service and workforce planning to meet health and social care needs associated with frailty.

Methods: The study will use a System Dynamics design to develop and test the simulation model.

Work packages comprise a scoping review, gathering of public and professional perspectives on service provision via a survey and stakeholder engagement activities, and analysis of linked health and social care data, all of which inform the simulation modelling work package and development of a workforce planning toolkit.

Timelines for delivery: The scoping review will be completed in year 1. Routine health and social care data specification and extraction will occur in year 1, as will service mapping and classification and survey preparation. Survey data collection and analysis will occur in year 2. Simulation modelling will commence in year 2, with validation, sensitivity analyses and scenario modelling in year 3.

Development of workforce guidelines and toolkit will occur in year 3 Stakeholder engagement, including patient public involvement, will run throughout the study, reviewing study results and informing development of the other work packages.

Anticipated impact & dissemination: This study will provide new, direct evidence about the impact of frailty on health and social care workforce requirements within the ageing population The improved understanding of workforce requirements offered by this study will inform workforce planning for frailty services across health and social care, ensuring future benefit for patients through provision of timely and appropriate care and a workforce planning toolkit to support local decision-making.

ELIGIBILITY:
Eligibility:

* Age 50yrs and above,
* contributing data to the North West London NHS Integrated Care System database

Exclusion:

*Age below 50yrs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age 50 and above
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Service use (for cohort analysis) | 2015-2022
  Use of primary, secondary, community, health and social care services

SECONDARY OUTCOMES:
Workforce provision of services to Adults living with Frailty | 2015-2022
  Information from cohort analysis, health and social care professionals survey and scoping review.

CONTACTS AND LOCATIONS:
Overall Officials: Bronagh M Walsh/Professor, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data dictionary; variables; types of data
Supporting Information: Study Protocol, CSR
Time Frame: Protocol - during study period Results and data - end of 2025
Access Criteria: Research Report to funder Published Papers
URL: https://fundingawards.nihr.ac.uk/award/NIHR134305

REFERENCES:
- See also: Funder website — https://fundingawards.nihr.ac.uk/award/NIHR134305